CLINICAL TRIAL: NCT00153257
Title: Comparison of the Prosthesis Ugytex by the Trans-obturator Approach and Anterior Colporrhaphy for the Surgical Treatment of Anterior Vaginal Wall Prolapse
Brief Title: Comparative Study of Mesh Versus No Mesh in Prolapse Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: DRRC (Unknown); Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P040306; CRC04001
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2019-11-21 (Actual); Status verified 2019-10

CONDITIONS: Vaginal Prolapse; Cystocele
MeSH Terms: conditions — Uterine Prolapse; Cystocele

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ugytex (Other): Anterior repair reinforced by a specially designed mesh: UgytexTM
  Interventions: Device: Ugytex
- No device (No Intervention): standard anterior colporrhaphy

INTERVENTIONS:
Device: Ugytex — Anterior repair reinforced by a specially designed mesh: UgytexTM
  Arms: Ugytex

SUMMARY:
Hypothesis / aims of study A RCT has shown that results of prolapse repair via vaginal approach could be improved when a polypropylene mesh is used as tissue support (1). However, non protected heavy-weight meshes were associated with a high rate of local complications such as vaginal erosions and dyspareunia (2). The aim of this multicentre study is to evaluate anatomical and functional results of an innovative low-weight polypropylene mesh protected by an absorbable hydrophilic film in the prolapse repair by vaginal route, in comparison by the standard anterior colporrhaphy.

Study design, materials and methods This study involves 15 centres in French Private or Public Hospital. Patients will be randomly allocated to be operated by a standard anterior colporrhaphy or by an anterior repair reinforced by a specially designed mesh: UgytexTM (Sofradim, France). Ugytex is a low-weight (38g/m²) and highly porous (average porosity: 89%, pores over 1.5mm) polypropylene monofilament mesh offering tissue ingrowth and connective differentiation for a stable and long-term support. The mesh is coated with a hydrophilic film composed of atelocollagen, polyethylene glycol and glycerol. The absorbable coating protects delicate pelvic viscera from the risk of acute inflammation during the healing's inflammatory peak. Prolapse severity will be evaluated using the POP-Q system. In order to evaluate the patient's quality of life, the validated PFDI and the PFIQ questionnaires will be used preoperatively and during follow-up (3), as well as a validated questionnaire on sexual problems. The difference on one-year cure rate should be 15% (80% for the anterior colporrhaphy and 95% for the mesh repair). Then the estimated number of patient is 97 in each arm.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 60 years-old
* Anterior vaginal wall prolapse of stage 2 or more (POP-Q system)
* Symptomatic prolapse
* Informed consent signature obtained

Exclusion Criteria:

* Patient not able to read French language
* Patient with a anterior prolapse of stage 1
* Urinary of vaginal infection
* Hepatopathy with ascitis
* Diabetes uncontrolled
* Treatment by corticosteroids
* Previous pelvic irradiation
* Intraoperative bladder injury

Min Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2005-04; Primary Completion 2010-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
number of anatomical recurrences of anterior vaginal wall prolapse of stage 2 or more (POP-Q system) | 1 year
  POP-Q score

SECONDARY OUTCOMES:
Perioperative and postoperative morbidity | 3 years
  Number of Major and minor complication
Functionnal results following intervention | 3 years
  Symptoms and quality of life questionnaires
Rate of local complications of prosthesis (vaginal erosion, prosthesis shrinkage) | 3 years
Post-operative sexuality | 3 years
  PISQ score

CONTACTS AND LOCATIONS:
Overall Officials: Hervé Fernandez, MD, Study Director — Hôpital Béclère, Clamart, France
Locations (1):
- Hôpital Carémeau, Nîmes, France

IPD SHARING:
Plan to Share IPD: No